CLINICAL TRIAL: NCT04128436
Title: The Effect of Early and Mid Luteal Blood Progesterone Levels on Ongoing Pregnancy Rates in IVF Cycles With Fresh Blastocyst Transfer
Brief Title: The Effect of Luteal Blood Progesterone Levels on Ongoing Pregnancy Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Anatolia IVF and Women's Health Center (Unknown)
Responsible Party: Principal Investigator, Sezcan Mumusoglu, Assistant Professor, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HU01
Record Dates: First submitted 2019-09-17; First posted 2019-10-16 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Luteal Phase Progesterone Levels
Keywords: luteal phase; progesterone; in vitro fertilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Progesterone levels (Other): Patients will be divided into groups according to quartiles (25/50/75) of progesterone levels. Optimal range of progesterone levels for ongoing pregnancy rate will be calculated.
  Interventions: Other: Taking blood samples for analyzing progesterone levels

INTERVENTIONS:
Other: Taking blood samples for analyzing progesterone levels — As part of standard in vitro fertilization treatment, Crinone gel will be used starting the next morning following the oocyte pick-up (OPU) as a luteal phase support. On the trigger day, on the day OPU+2/3 (early luteal phase) and on the embryo transfer day (OPU+5, mid luteal phase) blood samples will be taken from patients for evaluating the progesterone levels. Blood samples will be collected at the 6th hour following the morning dose of vaginal progesterone gel. No other intervention will be done to the patients.

SUMMARY:
Progesterone (P4) is essential for the secretory development of endometrium and the maintenance of early pregnancy. In the luteal phase following controlled ovarian stimulation in in vitro fertilization (IVF) treatment, P4 profile is completely different from natural cycles (Fauser, 2002).

Since the optimal luteal P4 levels are not well known, in normal IVF treatment a standard regime of exogenous P4 is given without considering the ovarian response for stimulation and the steroid levels in luteal phase. In 2005 Humaidan et al, showed that following the fresh embryo transfer, low luteal P4 levels (39 nmol/l) has a negative impact on ongoing pregnancy rates (Humaidan, 2005). In the following randomized controlled trials (RCTs), the use of exogenous human chorionic gonadotropin (hCG) after gonadotropin releasing hormone (GnRH) agonist trigger as a luteal phase support (Humaidan, 2010, 2013), the mid luteal P4 levels increased to 77-409 nmol/l and birth rates per transfer raised to %24.

In the light of these, it is essential that the progesterone levels in luteal phase is above the certain threshold for induction of the normal secretory development of endometrium following the IVF treatment and for the maintenance of pregnancy.

The implantation window is defined as that period when the uterus is receptive for implantation of the free-lying blastocyst. For maximal effectiveness of assisted reproductive technologies in women, it is important to know the optimal time for embryo transfer which implies a need to predict the period of uterine receptivity. Blood progesterone levels can be an indirect indication for implantation window and the embryo transfer timing.

In a recent study by Vuong et al., marked inter-personal variation in early luteal circulating P4 levels have been reported following the same hCG trigger dose; since a freeze-all policy was adopted in that study, the inter-personal variation during the early luteal phase was entirely caused by differences in endogenous P4 production from the CL (Vuong, et al., 2020). In this study, almost one in five patients had already experienced a peak P4 concentration on OPU+2 day to OPU+3 day, and only one in seven had maximal concentrations on OPU+6 day, showing that a total of 85% of women experienced their highest P4 concentration before the period in which the peak was expected to be reached during a natural menstrual cycle (Andersen, et al., 2020). It is noteworthy that more than 40% of patients had a >50% decrease in P4 concentration between OPU+4 day and OPU+6 day; although exogenous P4 supplementation in women undergoing IVF will ameliorate this drop-in serum P4 to some extent, these findings clearly highlight the requirement for studies examining how the probability of achieving pregnancy in fresh cycles is affected by the timing and magnitude of the reduction in P4 concentrations (Vuong, et al., 2020). Variations in endogenous production might, in theory, originate from differences in "quality" of the CL as seen during the natural cycle (Hull, et al., 1982) and/or differences in serum concentrations of hCG during the early luteal phase used for triggering (Vuong, et al., 2020b).

The aim of this study is two fold; i) to investigate the effect of early and mid luteal P4 levels on ongoing pregnancy rates and to determine the optimal luteal P4 levels in IVF cycles following the fresh blastocyst transfer in order to improve the reproductive outcomes, ii) to investigate the impact of serial P4 levels on OPU+3 and OPU+5 and delta P4 (ΔP4; as calculated by subtracting the P4 level on OPU+3 from the P4 level on OPU+5) on ongoing pregnancy rates.

DETAILED DESCRIPTION:
During Covid-19 pandemic we decided to make an interim analysis in March 2020.

Since the shut down of the IVF clinics due to Covid-19 pandemic was over, we restarted our routine IVF practice and hence restarted recruitment of patients for this study.

ELIGIBILITY:
Inclusion Criteria:

* Cycles induced with GnRH agonist or GnRH antagonist protocol
* BMI<35 kg/m
* Retrieval of 3 or more metaphase II oocytes, irrespective of ovarian reserve testing

Exclusion Criteria:

* Cycles triggered with GnRH agonist or dual trigger
* Circulating progesterone > 1.5ng/mL on the day of trigger
* Cleavage stage embryo transfer

Max Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 340 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rates | 27 months
  Clinically proven pregnancy more than 12 weeks of gestation

SECONDARY OUTCOMES:
Early luteal phase blood progesterone levels | 24 months
  Concentration of blood progesterone on the day of OPU+2/3
Mid luteal phase blood progesterone levels | 24 months
  Concentration of blood progesterone on the day of OPU+5/ embryo transfer day
Delta P4 | 24 months
  ΔP4; as calculated by subtracting the P4 level on OPU+3 from the P4 level on OPU+5.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Yaralı, Professor, Principal Investigator — Hacettepe University
Locations (3):
- Androfert, Campinas, São Paulo, Brazil
- Aarhus University, Aarhus, Denmark
- Hacettepe University School of Medicine, Department of Ob/Gyn, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Uyanik E, Mumusoglu S, Polat M, Yarali Ozbek I, Esteves SC, Humaidan P, Yarali H. A drop in serum progesterone from oocyte pick-up +3 days to +5 days in fresh blastocyst transfer, using hCG-trigger and standard luteal support, is associated with lower ongoing pregnancy rates. Hum Reprod. 2023 Feb 1;38(2):225-236. doi: 10.1093/humrep/deac255. PMID 36478179